CLINICAL TRIAL: NCT04756882
Title: Clinical Evaluation of the Efficacy OF Botulinum Toxin A for Improving Facial Scars (Randomized Clinical Trial )
Brief Title: Clinical Evaluation of the Efficacy OF Botulinum Toxin A for Improving Facial Scars
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Omnia Shetta, researcher, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Oshetta
Record Dates: First submitted 2021-02-07; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Hypertrophic Scarring
Keywords: Botulinum Toxin Type A; facial scarring; wound healing
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): 6 patients received 12.5 speywood unit/cm (SU/cm) Dysport intramuscular & intradermal injections, within the first 5 postoperative days of the trauma
  Interventions: Drug: AbobotulinumtoxinA 500 UNT
- control group (No Intervention): of 6 patients that acted as the control group and received no treatment

INTERVENTIONS:
Drug: AbobotulinumtoxinA 500 UNT — Anaerobic fermentation of the bacterium Clostridium botulinum produces botulinum toxin. A range of different C. Botulinum strains have been recognized; eight immunologically different serotypes (type A-H) are created and consist of botulinum neurotoxin complexed with a number of related proteins.
  Neurotoxin type A preparations are the most widely used for therapeutic application. There are currently three leading botulinum neurotoxin type A (BoNT/A) products on the market in the Western Hemisphere: onabotulinumtoxinA (ONA; Botox/Vistabel, Allergan Inc., Irvine, CA, USA), abobotulinum toxin A (ABO; Dysport/Ipsen Limited, Slough Berkshire, UK), and incobotulinum toxin A (INCO; Xeomin/Bocouture, Merz Pharmaceuticals GmbH, Frankfurt, Germany). In nature, BoNT-A is synthesized as macromolecular protein complexes
  Other Names: Dysport
  Arms: study group

SUMMARY:
Background: Scars widen when the overlying musculature pulls apart suture lines. Because Botulinum Toxin A (BTA) is known to prevent fibroblast proliferation and it also induces temporary muscle paralysis, the purpose of this current study is to evaluate the beneficial effects of Botulinum toxin type A (BTA) on scar formation.

Aim of this study: The aim of this study is to evaluate the efficacy and safety of early postoperative Botulinum Toxin type A (BTA) injection on improving vertical or oblique facial surgical scars.

Materials and methods: Patients with vertical or oblique forehead lacerations, treated by primary closure, will be enrolled in this study and randomized into two groups: One group (n =6) will receive BTA injection within 5 days of primary closure and the other group (n = 6) will receive no further treatment. Vancouver scar scale (VSS) Scores and wound width will be determined at the 1, 3 and 6 months follow-up visits, along with clinical photographs.

Results: Data will be collected, tabulated and statically analyzed. Key words: Botulinum Toxin Type A; facial scarring; wound healing; scar maturation

DETAILED DESCRIPTION:
1. All procedures were performed under local anesthesia in Oral and Maxillofacial Surgery Department, Alexandria University.
2. Using nonalcoholic solution after makeup removal, a single surgeon performed the procedures under complete aseptic technique (Lee, Min et al. 2018).
3. All patients wore a disposable cap to contain hair.
4. We examined before treatment: the facial anatomy, mimic muscular contraction, facial expression, and any pre-existing asymmetry(Wilson 2006).
5. Immediately after taking the photographs, both the length and width of the forehead wound were measured directly on the patients using a digital vernier caliper by a single plastic surgeon blinded to the study condition.
6. Pain at the injected sites was minimized before each injection by applying topical anesthetics and cold iced devices.
7. Micro fine 1.0 ml insulin syringes with a 29-G or 30-G needle were used.
8. The dosages of the preparations are related to biological activity and are given in biological units (U). The units are termed according to the manufacturer as Speywood U (SU) for Dysport
9. The drugs used were AboBotulinumToxin A Dysport (500 Speywood U) is to be reconstituted with 2.0 mL of sodium chloride 9 mg/mL (0.9%) injection solution. This results in a clear solution containing the 500 Speywood units of the active ingredient in a concentration of 250 units per 1.0 mL of the reconstituted solution. The reconstitution is to be performed in accordance with the rules of good clinical practice, particularly with respect to asepsis and within 15 day of reconstitutin.(Hexsel, Rutowitsch et al. 2009, Scaglione 2016, Lee, Min et al. 2018).
10. The total dose is approximately 105 SU.
11. The total dose is divieded into 75 SU injected by a (1-ml, , 30-gauge needle) insulin syringe along the scar length at the rate of approximately 12.5 SU (0.15 ml) per cm of wound length, in a linear pattern on either side of the wound. , with the needle prick positined approximately 5 mm from the edge of the wound, The injection was repeated every cm throughout the entire wound length and 30 SU are injected into frontalis muscle.(Wilson 2006, Hu, Zou et al. 2018, Kim, Lee et al. 2019)
12. Injections were determined by a skin marker and done under the supervision of a qualified licensed supervisor.
13. due to muscles contraction The injections were carried out on skin folds and are performed at different levels (intramuscular, subcutaneous, or intradermal) in more points for each region. The injections were administrated directly into the point of intense muscular contraction. On the other hand, where the contraction was weak, the injection was done at a deep or superficial intradermal level. Depth depends also on the effect we want to achieve: an extreme effect for intramuscular, a soft effect for subcutaneous or intradermal.(Iozzo, Tengattini et al. 2014)
14. To prevent eyebrow ptosis, the drugs were not injected around the supraorbital rim.(Kim, Lee et al. 2019).

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged from 18 to 40 years.

  * Patients free from any systemic disease.
  * Patients who understand verbal and written instructions

Exclusion Criteria:

* • Patients with horizontal forehead lacerations.

  * Patients suffering from complicated forehead lacerations that require grafting.
  * Patients with forehead burns.
  * Patients with neuromuscular disorders.
  * Patients with previous surgical or non-surgical intervention.
  * Patients allergic to drugs used in this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-05-18 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
change in wound width | baseline, 1st, 3rd, 6th months
  The mean width of the forehead wound of each group was measured be a digital vernier caliper for both the 1-month, 3-month and 6-month visits
change of vancouver scar scale | baseline, 1st, 3rd, 6th months
  The Vancouver scar scale (VSS) was assessed by two plastic surgeons in an independent, blinded fashion to quantify scar appearance at the 1-month, 3-month and 6-month visits

SECONDARY OUTCOMES:
color differences | baseline, 1st, 3rd, 6th months
  Quantified color differences between the scar and surrounding normal skin were measured and compared using the Commission International d'Eclairage (CIE) L*a*b* color coordinates for each patient. L*a*b* values of the region of interest were obtained using Adobe Photoshop 7.0 (Adobe Systems Incorporated, San Jose, CA.)

CONTACTS AND LOCATIONS:
Overall Officials: mahitab M soliman, phd, Study Director — Alexandria University
Locations (1):
- oral & maxillofacial surgery department ,faculty of dentistry, Alexandria university, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No